CLINICAL TRIAL: NCT05610813
Title: Multicentre, Randomized, Open-label Study to Prove an Additional Benefit of the Full-spectrum Cannabis Extract VER-01 Over Opioids in the Treatment of Patients With Chronic Non-specific Low Back Pain
Brief Title: Comparison of VER-01 to Opioids in Patients With Chronic Non-specific Low Back Pain
Acronym: ELEVATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertanical GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VER-CLBP-002
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Chronic Non-specific Low Back Pain
MeSH Terms: interventions — Opiate Substitution Treatment; Analgesics, Opioid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test intervention: VER-01 (Experimental): VER-01 will be administered twice daily to patients randomized to treatment arm VER-01.
  Interventions: Drug: VER-01
- Comparative intervention: Opioid therapy (with an authorised and marketed opioid, ATC code N02A) (Active Comparator): Opioids will be administered according to the SmPC to patients randomized to treatment arm opioid therapy.
  Interventions: Drug: Opioid therapy

INTERVENTIONS:
Drug: VER-01 — Standardized oleoresin of Cannabis sativa L. folium cum flore, THC-chemotype (cannabis leaves and - flowers), corresponding to 21 mg (-)-trans-Δ9-Tetra-hydrocannabinol (THC) per gram drug product
  Other Names: trans-Δ9-Tetra-hydrocannabinol (THC)
  Arms: Test intervention: VER-01
Drug: Opioid therapy — The patient-specific selection of the marketed opioid (based on standard of care and provided for this study) is at the discretion of the investigator and made at Visit 1, i.e., before randomization at Visit 2.
  Other Names: Opioids
  Arms: Comparative intervention: Opioid therapy (with an authorised and marketed opioid, ATC code N02A)

SUMMARY:
Randomized, open-label, parallel-group phase III trial to prove an additional benefit of the full-spectrum cannabis extract VER-01 over opioids in patients with chronic non-specific low back pain for whom drug treatment is indicated and previous optimized treatments with non-opioid analgesics have not led to sufficient pain relief or were unsuitable due to contraindications or intolerance.

DETAILED DESCRIPTION:
The test intervention VER-01 is a cannabis-based pain medication currently under clinical development that is expected to provide adequate pain relief while being better tolerated in long-term treatment compared to opioid analgesics. This study aims to demonstrate the superior tolerability, especially in terms of bowel function, of VER-01 compared to existing authorised and marketed opioid analgesics in patients with chronic non-specific low back pain. In addition, the safety and tolerability as well as the efficacy of VER-01 compared to opioid therapy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥18 years of age
2. Provision of informed consent form voluntarily signed and dated by the patient
3. For women of childbearing potential and men of reproductive potential: use of a reliable contraceptive method (Pearl index < 1) at least 1 month before the start of the study and willingness to use it during the study participation and 3 months after the last intake of the test or comparative intervention
4. Patient understands the local language and is willing and able to comply with scheduled visits, treatment plan, patient diary and other study related procedures throughout study participation
5. Chronic (for at least 3 months) non-specific pain in the lower back (between the 12th thoracic vertebra and lower gluteal folds). Non-specific pain refers to pain without a clear specific treatable cause.
6. Patients with indicated drug treatment where previous optimized treatments with non-opioid analgesics (including combinations) have not led to sufficient pain relief or were unsuitable due to contraindications or intolerance.
7. Low back pain intensity on average at least 4 points on an 11-point Numeric Rating Scale in the last 4 weeks prior visit 1
8. Ongoing non-drug pain therapy (physical or behavioral therapy) must have been stable for at least 2 weeks prior visit 1 and must be continued during the run-in phase
9. Ongoing additional analgesic treatment prior visit 1 must be continued during the run-in phase
10. Bowel Function Index total score of 28.8 or less at visit 1.

Exclusion Criteria:

1. Patients with a known history of alcohol/drug/medication abuse or dependency and previous or current use of methadone
2. Evidence of drugs of abuse or illegal drugs by urine drug test performed at visit 1
3. Known intolerance or hypersensitivity to ingredients of rescue medication, opioid therapy (assigned by the investigator) and/or VER-01
4. Participation in another clinical interventional study within the last 30 days prior screening visit (visit 1)
5. Occupational groups with primary activity of operating machinery and driving motor vehicles
6. Planned blood donation or planned donation or freezing of sperm or oocytes during study participation and 3 months after end of study participation
7. Pregnant or breastfeeding female patients
8. Patient is unable to provide written informed consent, in need for care, has a guardian/caretaker, is immobile, or is particularly vulnerable (e.g., imprisoned; institutionalised by a court or judicial authority; dependent or employed by the sponsor, an external service provider of the sponsor (involved in the conduct of the study), the investigator or the trial site)
9. Known use of opioid or cannabis-based treatments within 30 days before screening visit (visit 1)
10. Patients for whom cannabis or opioid therapy is not indicated, e.g., due to a history of non-response to opioid therapy or cannabis-based medicines in the treatment of chronic non-specific low back pain in the past.
11. Start of or planned non-drug pain therapy during run-in phase (physical or behavioral therapy)
12. Start or planned start of an additional analgesic treatment during run-in phase
13. Ongoing monoamine oxidase inhibitor therapy at screening visit (visit 1)
14. Patients with history of cancer in the last 5 years prior to screening visit (visit 1). Except for cutaneous basal cell or squamous cell cancer resolved by excision without recurrence and cervical cancer in situ resolved by excision with negative pap test.
15. Painful comorbidities which could interfere with the low back pain intensity assessment during the study
16. Known history of human immunodeficiency virus (HIV) infection
17. Severe forms of the following diseases: Anaemia, haematological / autoimmune / endocrine / renal / hepatic / respiratory / cardiovascular / neurological / gastrointestinal / symptomatic peripheral vascular diseases.
18. Cardiovascular event in the last three months before screening visit (visit 1)
19. Known uncontrolled hypertension (average systolic blood pressure ≥140 mmHg or average diastolic blood pressure

    ≥90 mmHg) and/or untreated hypothyroidism
20. Patients with Crigler-Najjar syndrome, Rotor syndrome and/or porphyria
21. History of major trauma or back surgery in the last 2 months prior to screening visit (visit 1)
22. Known history of or current severe psychiatric illness
23. Known history of or current severe depression (not due to chronic low back pain) (assessed by Patient Health Questionnaire - 9) and/or suicidal ideation (assessed by Columbia-Suicide Severity Rating Scale) at screening visit (visit 1)
24. Patients with severe respiratory depression
25. Patients with lung disease associated with impaired lung function (e.g., acute or severe bronchial asthma or hypercapnia/respiratory failure).
26. Patients with conditions of increased intracranial pressure due to head injury or disease of the brain.
27. Patients with existing or suspected paralytic ileus
28. Patients with intestinal obstruction due to intestinal paralysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Risk of developing constipation | 190 days
  Number and proportion of constipation responders at the end of treatment phase (Visit 9). A constipation responder is defined as a patient with
  1. a change from baseline (visit 2) in Bowel Function Index (BFI) total score of at least 15 points at Visit 9 and
  2. a BFI total score of more than 28.8 at Visit 9.

SECONDARY OUTCOMES:
Efficacy based on pain reduction | 190 days
  Number and percentage of 30% pain responders at study week 27 (last week of treatment phase) compared with the baseline score (study week -1)
Efficacy based on pain reduction in NE patients | 190 days
  Number and percentage of 30% pain responders in the subgroup of patients with a neuropathic pain component (painDETECT score >18) at study week 27 compared with the baseline score (study week -1)
Efficacy based on pain reduction and interference with sleep | 190 days
  Number and percentage of patients with a 30% improvement of the mean daily low back pain interference with sleep score evaluated on an 11-point Numeric Rating Scale (NRS) at study week 27 compared with the baseline score (study week -1)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Karst, Prof.Dr.med., Principal Investigator — Medizinische Hochschule Hannover (MHH)
Locations (2):
- Germany (2):
  - Rheumazentrum Prof. Dr. med. Gunther Neeck, Bad Doberan
  - Medizinische Hochschule Hannover (MHH), Hanover

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meissner W, Argoff C, Sator S, Schoder V, Karst M. VER-01 Shows Enhanced Gastrointestinal Tolerability, Superior Pain Relief, and Improved Sleep Quality Compared to Opioids in Treating Chronic Low Back Pain: A Randomized Phase 3 Clinical Trial. Pain Ther. 2025 Dec;14(6):1765-1782. doi: 10.1007/s40122-025-00773-z. Epub 2025 Sep 30. PMID 41028525